CLINICAL TRIAL: NCT05061563
Title: An Open-label, Non-randomized,Fixed-sequence Crossover Study to Investigate the Effects of a Proton Pump Inhibitor on the Pharmacokinetics of Elinzanetant (BAY 3427080) as Well as Assessment of the Absolute Bioavailability of Elinzanetant Using a Single Intravenous Microtracer Dose of [13C5]BAY 3427080 in Male and Female Healthy Participants
Brief Title: A Study to Learn How a Proton Pump Inhibitor Affects the Way Elinzanetant (BAY 3427080) Moves Into, Through and Out of the Body, and How Much of it Gets Absorbed by the Body When Taken as a Single and Small Radioactive Dose in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21772; 2021-002032-24 (EudraCT Number)
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men; Hot Flashes
Keywords: Hot flushes; Vasomotor symptoms; Elinzanetant; Drug-drug interaction; Proton pump inhibitor; Pharmcokinetics
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Hot Flashes | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): A single dose of elinzanetant and an additional IV (microtracer dose) of [13C5]BAY 3427080 will be administered.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Period 2 (Experimental): Once daily oral dose of esomeprazole and a single oral dose of elinzanetant will be administered.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Esomeprazole

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Elinzanetant given orally as single dose capsule and intravenous as single dose in Period 1. Elinzanetant given orally as single dose capsule in Period 2.
  Other Names: NT-814
Drug: Esomeprazole — Esomeprazole given orally once daily for 5 days in Period 2.
  Arms: Period 2

SUMMARY:
Researchers are looking for a better way to treat people who have vasomotor symptoms (VMS). VMS such as hot flashes are caused by hormonal changes occurring during menopausal transition when women may have also changes in their monthly cycles.

The study treatment, elinzanetant (BAY3427080), was developed to work by blocking neurokinin receptors from working. These receptors can cause changes in the body which can affect hormone levels in men and women.

Acid is created by the stomach to help break down and digest food. A type of treatment for overly production of acid by the stomach are called proton pump inhibitors which are currently available for people who have stomach and digestion problems. Proton pump inhibitors work by lowering the amount of acid created by the stomach. In this study, the researchers want to learn about elinzanetant oral bioavailability when taken with a proton pump inhibitor called esomeprazole. They want to learn if taking these drugs together affects the oral bioavailability.

The researchers will study how esomeprazole affects the way elinzanetant moves into, through, and out of the body. To do this, the doctors and their team will take blood samples from the participants. These samples will be used to measure the levels of elinzanetant in the participants' blood when it is taken with and without esomeprazole.

This study will include healthy adult participants.

There will be 2 periods in this study. It is planned that all of the participants will take part in both periods. During Period 1, the participants will take elinzanetant 1 time as a capsule by mouth. The participants will also receive a very small amount of radioactive elinzanetant, also called a microtracer, given through needle in a vein. During Period 2, the participants will take esomeprazole once a day for 5 days as tablets by mouth. On the last day, the participants will also take elinzanetant 1 time as a capsule by mouth.

During this study, the participants will visit the study site 3 times. The participants will stay at the study site for 9 days in Period 1 and for 12 days in Period 2. Each participant will be in the study for up to 9 weeks.

During the study, the doctors will take urine samples. They will also ask the participants about any medications they have been taking, and what adverse events they are having. An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight of at least 50 kg and body mass index (BMI) within the range of 18.0 to 30.0 kg/m^2 (inclusive).
* Male and female Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * Male participants: Male participants of reproductive potential must agree to use a condom (with or without spermicide) when sexually active. This applies for the time period between the signing of the informed consent form (ICF) until 5 days after the last dose of study intervention. Female partners of childbearing potential of male participants do not need to follow special precautions.
  * Female participants: Women of childbearing potential will have to use highly effective non-hormonal contraception when having sexual intercourse with a male partner from signing the ICF until 5 days after last dose of the study drug.
  * Women of non-childbearing potential are not required to use contraception. Non-childbearing potential is defined as
* Postmenopausal state confirmed by follicle stimulating hormone (FSH) level >33.4 U/L, or above reference range from the local laboratory, or
* Surgically sterilized by bilateral tubal ligation, bilateral oophorectomy with or without hysterectomy, or hysterectomy documented by medical report verification.

Exclusion Criteria:

* Any clinically relevant abnormal findings in medical history and physical examination which in the opinion of the investigators, may put the participant at risk because of his/her participation in the trial or provide difficulties in interpreting the trial data.
* History or evidence of any clinically relevant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other clinically relevant disease, as judged by the investigator.
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal.
* Any medical disorder, condition or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator.
* Known hypersensitivity to the study interventions (active substances, or excipients of the preparations).
* Known severe allergies e.g., allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids, urticaria or significant non-allergic drug reactions.
* Relevant diseases within the last 4 weeks prior to the first study intervention administration.
* Febrile illness within 4 weeks before first study intervention administration.
* Contraindications for the use of esomeprazole, especially known hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency
* Use of drugs which may affect absorption (e.g. loperamide, metoclopramide) within 1 week before first study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Area under the concentration vs. time curve from zero to infinity after single (first) dose (AUC) of elinzanetant without concomitant administration of esomeprazole. | Period 1: Predose, Day 1 to Day 8.
  (AUC(0-tlast) will be used as main parameter if AUC cannot be calculated.)
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of elinzanetant without concomitant administration of esomeprazole. | Period 1: Predose, Day 1 to Day 8.
Area under the concentration vs. time curve from zero to infinity after single (first) dose (AUC) of elinzanetant with concomitant administration of esomeprazole. | Period 2: Predose, Day 1 to Day 8.
  (AUC(0-tlast) will be used as main parameter if AUC cannot be calculated.)
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of elinzanetant with concomitant administration of esomeprazole. | Period 2: Predose, Day 1 to Day 8.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs). | After first application of intervention up to 21 days after last dosing.
Absolute bioavailability (F) of Elinzanetant. | Period 1 : Predose, Day 1 to Day 8.

CONTACTS AND LOCATIONS:
Locations (1):
- PRAHealthSciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.